# Administrative information:

| Sponsor name | Diakonhjemmet Hospital |
|---|---|
| Sponsor address | Postboks 23 Vinderen<br>0319 Oslo<br>Norway |
| REC no | 477746 |
| Trial title | Happy Hands – an e-self-management intervention for people with hand osteoarthritis |
| PVO no | 00660 |
| Trial registration number | NCT05568875 https://clinicaltrials.gov/study/NCT05568875?term=NCT05568875&rank=1 |

# SAP and protocol version:

| SAP version and date: | This SAP is version 1.0, 21.03.2025 |
|-----------------------|-------------------------------------|

# SAP revision history:

| SAP<br>version | Section number changed | Description and reason for change | Date changed |
|---|---|---|---|
| version | changeu | | |
| 1.0 | NA | Original file | 21.03.2025 |
| 1.0 | 10. | Ong.mar me | 21.03.2023 |
| NA | | | |

# SIGNATURE PAGE

# PRINCIPAL/COORDINATING INVESTIGATOR:

Anne Therese Tveter, PhD Senior researcher | Professor Health Service Research and Innovation Unit (EHI) Diakonhjemmet Hospital

| Anne Therese Tveter | 21.03.2025 |
|---|---|
| Signature | Date (dd/mmm/yyyy) |
| DATA ANALYST: | |
| Joseph Sexton, PhD<br>Senior researcher<br>Diakonhjemmet Hospital | |
| forSV | |
| (" | 02.04.2025 |
| Signature | Date (dd/mmm/vvvv) |

# **ABBREVIATIONS**

| AE | Adverse event |
|---|---|
| BMI | Body Mass Index |
| CONSORT | Consolidated Standards of Reporting Trials |
| eHEALS | The eHealth Literacy Scale |
| EQ-5D-5L | EuroQol |
| НОА | Hand osteoarthritis |
| ICER | incremental cost-effectiveness ratio |
| MAP-Hand | Measure of Activity Performance of the Hand |
| NSAIDs | Non-Steroid Anti-Inflammatory Drugs |
| NRS | Numeric rating scale |
| OA | Osteoarthritis |
| OMERACT | Outcome Measures in Rheumatology (Outcome Measures in Rheumatoid Arthritis Clinical Trials) |
| OARSI | Osteoarthritis Research Society International |
| QALY | Quality-adjusted life year |
| RCT | Randomized controlled trial |
| REK | Regional committee |
| SAE | Serious adverse event |
| SUS | System Usability Scale |
| TSD | Services for sensitive data (Tjeneste for sensitive data) |

# TABLE OF CONTENTS

| 1. | INT | TRODUCTION | 5 |
|---|---|---|---|
| | 1.1 | Background and rationale | |
| | 1.2 | Trial Objectives | 5 |
| | 1.2.1 | Primary Objective | 5 |
| | 1.2.2 | Secondary Objectives | 5 |
| | 1.2.3 | Exploratory Objectives | 6 |
| 2. | TRI | AL METHODS | 7 |
| | 2.1 | Trial Design | 7 |
| | 2.2 | Randomization | 7 |
| | 2.3 | Sample size | 8 |
| | 2.4 | Statistical Framework | 8 |
| | 2.4.1 | Hypothesis Test | 8 |
| | 2.4.2 | Secondary hypotheses | 9 |
| | 2.4.3 | Other objectives | 11 |
| | 2.4.4 | Decision Rule | |
| | 2.5 | Statistical Interim Analyses and Stopping Guidance | |
| | 2.6 | Timing of Final Analysis | |
| | 2.7 | Timing of Outcome Assessments | |
| 3. | STATISTICAL PRINCIPLES | | |
| | 3.1 | Adherence and Protocol Deviations | |
| | 3.1.1 | Adherence to Allocated Treatment | 13 |
| | 3.1.2 | Protocol Deviations | 13 |
| | 3.2 | Analysis Populations | |
| 4. | TRI | AL POPULATION | 14 |
| | 4.1 | Screening Data, Eligibility and Recruitment | 14 |
| | 4.2 | Withdrawal/Follow-up | 16 |
| | 4.3 | Baseline Patient Characteristics | 16 |
| 5. | AN | ALYSIS | 16 |
| | 5.1 | Outcome Definitions | 16 |
| | 5.1.1 | General Definitions and Derived Variables | 16 |
| | 5.1.2 | Primary Outcome Definitions | 18 |
| | 5.1.3 | Secondary Outcomes Definitions | 19 |
| | 5.1.4 | Overview of Outcomes | 19 |
| | 5.2 | Analysis Methods | |
| | 5.2.1 | Primary Outcome | |
| | 5.2.2 | Secondary Outcomes | |
| | 5.2.3 | Additional Analyses | |
| 6. | | FETY ANALYSES | |
| ٥. | 6.1 | Adverse Events/Safety | |
| 7. | | ATISTICAL SOFTWARE | |
| 8. | | HICS 26 | 20 |
| 9. | | FERENCES | 26 |

## 1. Introduction

## 1.1 Background and rationale

Osteoarthritis (OA) is a prominent cause of years lived with disability worldwide [1]. The hand is one of the most commonly affected sites [2] with a lifetime risk of 50% in women and 25% in men for developing hand OA (HOA) [3]. There are no disease-modifying drugs that can cure HOA. Patient education, hand exercises, and assistive devices are the core treatments, while Non-Steroid Anti-Inflammatory Drugs (NSAIDs) can be used for a limited duration to relieve symptoms [4]. Surgery should only be considered if other treatment modalities are ineffective [4]. Core treatment should primarily be provided in primary healthcare, however, research shows that the quality-of-care of OA-services in general is sub-optimal [5], and in particular for people with HOA [6,7].

The use of eHealth is highlighted for self-management and better exploitation of healthcare resources [8]. An observational study suggests that digital delivery of core treatment could be a viable option in people with HOA [9], however, large methodologically sound trials of effect and cost-effectiveness are lacking [10].

In 2020, development of the Happy Hands app was initiated at Diakonhjemmet Hospital, Norway [11], with an overarching goal of delivering a standalone intervention that supports and empowers people with HOA to self-manage their disease, regardless of where they reside [11]. Feasibility of the app has been tested in 71 patients with HOA with promising results [12], and there is now a need to test the app in an RCT to assess the effect and cost-effectiveness.

## 1.2 Trial Objectives

### 1.2.1 Primary Objective

The primary objective of this study is to assess whether a 12-week self-management intervention delivered through the Happy Hands app in addition to usual care is more effective compared to usual care alone in patients with HOA with regards to the **probability of OMERACT/OARSI response** at **3 months**.

# 1.2.2 Secondary Objectives

Key secondary objectives are:

- To assess whether a 12-week self-management intervention delivered through the Happy Hands app in addition to usual care is more effective compared to usual care alone in patients with HOA with regards to the probability of OMERACT/OARSI response at 6 months.
- To assess whether a 12-week self-management intervention delivered through the Happy Hands app in addition to usual care is cost-effective compared to usual care alone in patients with HOA at 6 months.

- To assess whether a 12-week self-management intervention delivered through the Happy Hands app in addition to usual care is more effective than to usual care alone in patients with HOA with regards to change in pain at 3 months.
- To assess whether a 12-week self-management intervention delivered through the Happy Hands app in addition to usual care is more effective than to usual care alone in patients with HOA with regards to **change in hand function** at **3 months.**

#### Other secondary objectives are:

- To assess whether a 12-week self-management intervention delivered through the Happy Hands app in addition to usual care is more effective than to usual care alone in patients with HOA with regards to change in grip strength at 3 months.
- To assess whether a 12-week self-management intervention delivered through the Happy Hands app in addition to usual care is more effective than to usual care alone in patients with HOA with regards to change in quality of care at 3 months.
- To assess whether a 12-week self-management intervention delivered through the Happy Hands app in addition to usual care is more effective than to usual care alone in patients with HOA with regards to change in disease activity at 3 months.
- To assess whether a 12-week self-management intervention delivered through the Happy Hands app in addition to usual care is more effective than to usual care alone in patients with HOA with regards to **change in pain** at **6 months**.
- To assess whether a 12-week self-management intervention delivered through the Happy Hands app in addition to usual care is more effective than to usual care alone in patients with HOA with regards to change in hand function at 6 months.
- To assess whether a 12-week self-management intervention delivered through the Happy Hands app in addition to usual care is more effective than to usual care alone in patients with HOA with regards to change in grip strength at 6 months.
- To assess whether a 12-week self-management intervention delivered through the Happy Hands app in addition to usual care is more effective than to usual care alone in patients with HOA with regards to change in quality of care at 6 months.
- To assess whether a 12-week self-management intervention delivered through the Happy Hands app in addition to usual care is more effective than to usual care alone in patients with HOA with regards to change in disease activity at 6 months.

## 1.2.3 Exploratory Objectives

- To assess the adherence, satisfaction and usability of the Happy Hands
- To identify factors associated with being an OMERACT/OARSI responder at 3 and 6 months

 To identify factors associated with adherence to the self-management intervention delivered through the Happy Hands app.

#### 2. Trial Methods

### 2.1 Trial Design

The Happy Hands study is designed as a pragmatic, open-labelled, 2-armed, randomized, controlled, multicenter, single-country trial. Participants are randomly allocated to either usual care (control group) or usual care combined with use of the Happy Hands app across a 12-weeks period (intervention group).

## 2.2 Randomization

Eligible patients are allocated in a 1:1 ratio between control group and intervention group through electronic questionnaires using Nettskjema. Through a build-in Javascript based randomization module, participants are randomly allocated by being forwarded from one questionnaire (the consent form) to one of two baseline questionnaires; one for the control group and one for the intervention group. These questionnaires are identical except for some questions being omitted in the baseline questionnaire for the intervention group as these are answered in the app. After answering the baseline questionnaire, the participants are forwarded to yet another questionnaire, informing them about group allocation. The intervention group is forwarded to yet another questionnaire where they are provided with the link to download the Happy Hands app. Patients (and healthcare provider) are blinded to group allocation until the patient has answered the baseline questionnaire, after that there is no possibility to blind neither patient nor healthcare provider.

The randomization is stratified by recruitment site. A total of 20 sites will recruit participants, thus, altogether 20 identical consent forms, and 20 identical baseline questionnaires for the control group and the intervention group, respectively, have been generated in Nettskjema. Examples of the randomization procedure is provided in Figure 1A and 1B.



Figure 1A: Example of randomization process for recruitment site 1



Figure 1B: Example of randomization process for recruitment site 2.

The group allocation questionnaires and the questionnaire containing link to downloading of the app are the same for all recruitment sites as the randomization has been conducted prior to being forwarded to these questionnaires.

# 2.3 Sample size

The sample size is calculated based on the primary outcome (proportion of OMERACT-OARSI responders) measured at 3 months. An OMERACT-OARSI responder rate between 26-46% is previously shown in hand exercise groups compared to 6-24% in usual care groups [13,14]. The between-group difference in primary outcome is estimated to 20% [15]. To account for multiple testing (primary and key secondary hypotheses), we will use a significance level of 1%, and 90% power. With a between-group difference of 20% and a usual care responder rate of 20%, we need to include 150 patients in each group. To account for a possible drop-out rate of 25% due to the digital nature of the study, a total of 376 patients are needed.

More detailed information is available in the study protocol [12].

# 2.4 Statistical Framework

## 2.4.1 Hypothesis Test

This trial is designed to assess if using the Happy Hands app in addition to usual care is superior to usual care alone with regards to probability of OMERACT/OARSI response at 3 months.

 The primary null hypothesis posits that there is no difference in probability of OMERACT/OARSI response between Happy Hands in addition to usual care compared to usual care alone at 3 months.

The primary alternative hypothesis is that using the Happy Hands app in addition to usual
care is superior to usual care alone with regards to probability of OMERACT/OARSI response
at 3 months.

#### 2.4.2 Secondary hypotheses

## Key secondary hypotheses:

- a) To assess the effect of using the Happy Hands app in addition to usual care compared to usual care only with regards to probability of OMERACT-OARSI response at 6 months.
  - The null hypothesis posits that there is no difference in probability of OMERACT/OARSI response between using Happy Hands in addition to usual care compared to usual care alone at 6 months.
  - The alternative hypothesis is that using Happy Hands in addition to usual care is superior to usual care alone with regards to probability of OMERACT/OARSI response at 6 months.
- b) To assess the cost-effectiveness of using the Happy Hands app in addition to usual care compared to usual care alone at 6 months.
  - The null hypothesis is that the Happy Hands intervention is not cost-effective compared to usual care alone at 6 months.
  - The alternative hypothesis is that using the Happy Hands app is cost-effective compared to usual care alone at 6 months.
- c) To assess the effect of using the Happy in addition to usual care compared to usual care alone on the change in pain from baseline to 3 months.
  - The null hypothesis is that there is no difference in change in pain from baseline to 3 months follow-up between using Happy Hands in addition to usual care compared to usual care alone.
  - The alternative hypothesis is that using the Happy Hands app in addition to usual care in more effective regarding change in pain from baseline to 3 months follow-up compared to usual care alone.
- d) To assess the effect of using the Happy in addition to usual care compared to usual care alone on the change in function from baseline to 3 months.
  - The null hypothesis is that there is no difference in change in function from baseline to 3 months follow-up between using Happy Hands in addition to usual care compared to usual care alone.
  - The alternative hypothesis is that using the Happy Hands app in addition to usual care in more effective regarding change in function from baseline to 3 months follow-up compared to usual care alone.

# Additional secondary hypotheses:

a) To assess the effect of using the Happy in addition to usual care compared to usual care alone on the change in grip strength from baseline to 3 months.

- The null hypothesis is that there is no difference in change in grip strength from baseline to 3 months follow-up between using Happy Hands in addition to usual care compared to usual care alone.
- The alternative hypothesis is that using the Happy Hands app in addition to usual care in more effective regarding change in grip strength from baseline to 3 months follow-up compared to usual care alone.
- b) To assess the effect of using the Happy in addition to usual care compared to usual care alone on the change in disease activity from baseline to 3 months.
  - The null hypothesis is that there is no difference in change in disease activity from baseline to 3 months follow-up between using Happy Hands in addition to usual care compared to usual care alone.
  - The alternative hypothesis is that using the Happy Hands app in addition to usual care in more effective regarding change in disease activity from baseline to 3 months follow-up compared to usual care alone.
- c) To assess the effect of using the Happy in addition to usual care compared to usual care alone on the change in quality of care from baseline to 3 months.
  - The null hypothesis is that there is no difference in change in quality of care from baseline to 3 months follow-up between using Happy Hands in addition to usual care compared to usual care alone.
  - The alternative hypothesis is that using the Happy Hands app in addition to usual care in more effective regarding change in quality of care from baseline to 3 months follow-up compared to usual care alone.
- d) To assess the effect of using the Happy in addition to usual care compared to usual care alone on the change in pain from baseline to 6 months.
  - The null hypothesis is that there is no difference in change in pain from baseline to 6 months follow-up between using Happy Hands in addition to usual care compared to usual care alone.
  - The alternative hypothesis is that using the Happy Hands app in addition to usual care in more effective regarding change in pain from baseline to 6 months follow-up compared to usual care alone.
- e) To assess the effect of using the Happy in addition to usual care compared to usual care alone on the change in function from baseline to 6 months.
  - The null hypothesis is that there is no difference in change in function from baseline to 6 months follow-up between using Happy Hands in addition to usual care compared to usual care alone.
  - The alternative hypothesis is that using the Happy Hands app in addition to usual care in more effective regarding change in function from baseline to 6 months follow-up compared to usual care alone.
- f) To assess the effect of using the Happy in addition to usual care compared to usual care alone on the change in grip strength from baseline to 6 months.
  - The null hypothesis is that there is no difference in change in grip strength from baseline to 6 months follow-up between using Happy Hands in addition to usual care compared to usual care alone.

- The alternative hypothesis is that using the Happy Hands app in addition to usual care in more effective regarding change in grip strength from baseline to 6 months follow-up compared to usual care alone.
- g) To assess the effect of using the Happy in addition to usual care compared to usual care alone on the change in disease activity from baseline to 6 months.
  - The null hypothesis is that there is no difference in change in disease activity from baseline to 6 months follow-up between using Happy Hands in addition to usual care compared to usual care alone.
  - The alternative hypothesis is that using the Happy Hands app in addition to usual care in more effective regarding change in disease activity from baseline to 6 months follow-up compared to usual care alone.
- h) To assess the effect of using the Happy in addition to usual care compared to usual care alone on the change in quality of care from baseline to 6 months.
  - The null hypothesis is that there is no difference in change in quality of care from baseline to 6 months follow-up between using Happy Hands in addition to usual care compared to usual care alone.
  - The alternative hypothesis is that using the Happy Hands app in addition to usual care in more effective regarding change in quality of care from baseline to 6 months follow-up compared to usual care alone.

## 2.4.3 Other objectives

Other objectives are considered to be supportive or exploratory, thus, they are not subject to hypothesis testing.

## 2.4.4 Decision Rule

For the primary outcome, superiority of probability of OMERACT/OARSI response is claimed if the null hypothesis is rejected at the significance level (alpha) of 0.01 (Bonferroni corrected due to multiple testing of one primary and four key secondary hypotheses; 0.05/5= 0.01. The result is deemed clinically relevant if the lower limit of the 95% confidence interval is more than 20% (see figure 2).

A significance level of <0.01 will also be used for the four key secondary hypotheses due to multiple testing.

For the additional secondary outcomes, multiple testing adjustment will not be carried out. The listed hypotheses will be assessed by their (unadjusted) p-values though no formal acceptance/rejection of these hypotheses will be done.

The intervention will be considered cost-effective if the incremental cost effectiveness ratio is below the threshold for cost-effectiveness, recommended in Norway. In the health economic evaluation, we will not consider p-values or confidence intervals for the ICER but instead plot bootstrapped ICERs on the cost-effectiveness plane and calculate a cost-effectiveness acceptability curve [16].



Figure 2: Visualization of superiority and clinically relevant difference.

# 2.5 Statistical Interim Analyses and Stopping Guidance

There will be no interim analyses in this trial.

# 2.6 Timing of Final Analysis

The main analysis is planned when all patients are finished with the data collection, all data have been entered, verified and validated and the primary database has been locked.

# 2.7 Timing of Outcome Assessments

Outcomes are assessed at baseline, 3 and 6 months. In addition, the intervention group will answer questionnaires as part of the Happy Hands app at a monthly basis and after each exercise session.

| Visit Label | Target Day | Definition (Day window) |
|---|---|---|
| T0. Consent | The day they consult a healthcare provider at one of the recruitment sites | Day 0 |
| T0. Randomization | After receiving information about the study, the participants are asked to sign a digital consent, thereafter the participants are randomly allocated to two groups based | Day 0 |

| | on baseline questionnaire (see section 2.2.) | |
|---|---|---|
| TO. Baseline | Day 0 Baseline assessment | Day 0 |
| T3. 3-months follow-up | Day 90 Follow-up (digital/face-<br>to-face) | Day 90 +/- 45 |
| T6. 6-months follow-up | Day 180 Follow-up (digital) | Day 180 +/- 45 |

# 3. Statistical Principles

#### 3.1 Adherence and Protocol Deviations

# 3.1.1 Adherence to Allocated Treatment

#### e-self-management intervention:

Adherence will be evaluated by tracking the number of exercise and informational videos viewed, as well as the number of quizzes completed each week. Each time a participant watches a video or submits quiz answers; this activity will be recorded in Nettskjema. Participants will also document each instance of exercise completion in the app. Recognizing that not all participants will view the same exercise videos multiple times, adherence to the exercise regimen will be based on self-reported exercise completion. As there is no consensus regarding what constitute adequate adherence to hand exercises, the American College of Sports Medicine guidelines will be used [17]. Adherence to the exercise program will be considered adequate if participants compete ≥2 exercise sessions per week for a duration of least 8 weeks (67%)[18]. Adherence to information videos and quizzes will be deemed adequate if participants have watched 19 of 26 videos and completed 9 of 12 quizzes, corresponding to approximately 75% utilization.

#### **Usual care:**

Usual care will vary between the different recruitment sites, from nothing to a single consultation, information courses or adaptation of orthosis. Thus, all participants are considered to have received usual care.

## 3.1.2 Protocol Deviations

Not all recruitment sites have the possibility to summon the participants for a face-to-face follow-up consultation. Thus, there will be a deviation from the protocol regarding the assessment of follow-up grip strength.

# 3.2 Analysis Populations

The Enrolled set will include all patients who have provided informed consent, have been included into the study data base, randomly assigned to one of the two groups and completed the baseline questionnaire.

The Full Analysis Set will be the same as the Enrolled set as the different questionnaires are linked together at baseline, thus, the patients will answer both consent, baseline questionnaire and be randomly allocated in one action.

The Per protocol set will include those who are deemed adherent based on the number of exercise session they have conducted and the number of informational videos they have seen.

# 4. Trial Population

## 4.1 Screening Data, Eligibility and Recruitment

The total number of screened patients and reasons for not entering the trial will be summarised and tabulated.

A CONSORT flow diagram (Figure 3) will be used to summarise the number of patients who were:

- · assessed for eligibility at screening
- eligible at screening
- ineligible at screening
- eligible and randomised
- eligible but not randomised
- · received the randomised allocation
- lost to follow-up 3 months
- lost to follow-up 6 months

Reasons will be provided where possible.



# 4.2 Withdrawal/Follow-up

The status of eligible and randomised patients at trial end will be tabulated by group according to

- withdrawn consent
- lost to follow-up

This will be presented in the CONSORT diagram.

## 4.3 Baseline Patient Characteristics

The patient demographics and baseline characteristics to be summarised include age, gender, living arrangement, education, occupational status, smoking, height and weight (calculated to BMI), most painful hand, other painful joints, previous treatment including surgery, medication, comorbidities, (e)Health literacy, joint mobility, pain at rest and in activity, disease activity, hand function, quality of care, health-related quality of life, motivation for exercising, grip strength.

Patient demographics and baseline characteristics will be summarised by randomised treatment arm and overall using descriptive statistics (mean, standard deviation, median, 25/75 percentiles) for continuous variables, and number and percentages for categorical variables. Any clinically important imbalance between the treatment groups will be noted.

# 5. Analysis

## 5.1 Outcome Definitions

### 5.1.1 General Definitions and Derived Variables

### 5.1.1.1 Age

Reported as age in years

## 5.1.1.2 Gender

Reported as male/ female/ other.

# 5.1.1.3 Living arrangements

Reported as living alone / living together with someone.

## 5.1.1.4 Education

Reported as elementary school / high school / college, university less than 4 years / college, university 4 years or more. Will be dichotomized into less than (elementary school/ high school) or more than (college, university) 12 years.

#### 5.1.1.5 Occupation status

Reported as working fulltime / working parttime / fulltime sick leave / parttime sick leave / retired / disability benefit / work assessment allowance / seeking work / unpaid, staying at home /student. Will be dichotomized to working/ not working.

#### 5.1.1.6 Smoking

Reported as smoking/ smoking previously/ not smoking.

#### 5.1.1.7 Height and weight (Body mass index, BMI)

Reported as body height (cm) and body weight (kg). Calculated as BMI = Body weight in kilograms divided by the square of the height in meters.

#### 5.1.1.8 Most troublesome joint

Reported as left hand/ right hand/ both hands/ none of the hands.

#### 5.1.1.9 Other troublesome joints

Reported as right hip/ left hip/ right knee/ left knee/ right ankle or foot/ left ankle or foot. Will be summarized into number of other troublesome joints (0-6)

#### 5.1.1.10 Previous treatment

Reported as having received previous treatment (yes/no) and a description of the treatment if reporting yes. Additionally, reported as previously having hand surgery (yes/no), and if yes, with hand (right/left/both).

#### 5.1.1.11 Medication

Reported as using medication due to hand OA (yes/no), with description of type and dose if answering yes.

### 5.1.1.12 Comorbidities

Reported as any problems affecting health (yes/no) for the following reasons: high blood pressure/ angina, infarction, other heart disease/ asthma, bronchitis, other lung disease/ allergy, eczema/ sciatic pain/ stroke, cerebral haemorrhage/ cancer/ neurological disease/ diabetes/ metabolic disease/ mental disease/ kidney disease/ liver disease/ ulcer, other stomach disease/ anaemia. Summarized as having comorbidity (yes/no), and number of comorbidities (0-15).

#### 5.1.1.13 (e)Health literacy

Measured by eHEALS [19,20], consisting of eight statements answered on 5-point scale (from "totally agree" to "totally disagree") with a total score ranging from 8 to 40 (higher score representing higher health literacy). Additionally, the participants are asked about their knowledge/experience with using technology and digital services like smartphone, tablets, apps, video consultation, and digital services (Helsenorge.no). The knowledge/experience with using measured on a 5-point scale (very poorly to very good) with an additional alternative of 'never tried'

## 5.1.1.14 Joint mobility

Measured using a numeric rating scale (NRS) from 0 to 10 with 0 being very good joint mobility. Reported separately for left and right hand. In baseline, 3- and 6-month questionnaires, the

participants are asked to rate their pain the last week. In the Happy Hands app, the participants are asked to rate their pain after exercising.

#### 5.1.1.15 Pain

Measured using an NRS from 0 to 10 with 0 being no pain. Reported separately for right and left hand at rest and in activity. In baseline, 3- and 6-month questionnaires, the participants are asked to rate their pain the last week. In the Happy Hands app, the participants are asked to rate their pain after exercising.

#### 5.1.1.16 Disease activity

Measured using an NRS from 0 to 10 with 0 being no disease activity.

## 5.1.1.17 Hand function

Measured by the Measure of Activity of the Hand (MAP-Hand) questionnaire, containing 18 questions about problems with different activities (no problems/ some problems/ large problems /cannot perform). A mean score (from 1 to 4 with 1 being no problems) is calculated from the answers, with at least 15 of 18 items having to be answered for a valid score [21].

#### 5.1.1.18 Quality of care

Measured by a modified version of the OsteoArthritis Quality Indicator questionnaire v2 [22], modified to hand OA. Containing 20 items related to treatment recommendations for hand OA, answered with yes/no/not relevant, do not have pain, do not remember. Scored as a pass rate (0-100%, with 100% being best quality of care), calculated as the number of yes-answers, divided by the total number of yes- and no-answers.

## 5.1.1.19 Health-related quality of life

Measured by EuroQol EQ-5D-5L [23], five items (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) scored at a 5-level scale ("no problems" to "unable to do"), calculated as a utility index 0-1, 1= best health-related quality of life. Visual analogue scale (EQ VAS), 0-100, 100= perfect health.

### 5.1.1.20 Grip strength

Maximum grip strength measured as the mean of two measures for left and right hand separately, using the JAMAR dynamometer. Grip strength is given in kg.

### 5.1.1.21 Motivation for exercising

Reported on an NRS from 0 to 10 with 0 being no motivation.

#### 5.1.1.22 Costs

Costs connected to patient care pathways will be self-reported by the patient using open-ended questions.

# 5.1.2 Primary Outcome Definitions

The primary outcome will be defined as OMERACT/OARSI responder [24], which is a composite index reported as a single variable (yes/no) based on one of the two following criteria:

Statistical Analysis Plan Happy Hands Diakonhjemmet Hospital

- High improvement on pain or function
  - $\circ$  ≥50% improvement + absolute change of ≥2 points in pain (NRS 0-10, 0=no pain), OR
  - ≥50% improvement + absolute change of ≥0.6 point in hand function (MAP-Hand 1-4, 1=no disability)
- Improvement in at least two of the three following
  - ≥20% improvement + absolute change of ≥1 points in pain (NRS 0-10, 0=no pain)
  - $\circ$  ≥20% improvement + absolute change of ≥0.3 point in hand function (MAP-Hand 1-4, 1=no disability)
  - ≥20% improvement + absolute change of ≥1 points in disease activity (NRS 0-10,
     0=no disease activity)

# 5.1.3 Secondary Outcomes Definitions

Secondary outcomes are listed in Table 1.

For assessment of cost-effectiveness, we will use healthcare costs (as listed under Costs in Table 1) and scores from EQ-5D-5L calculated into a utility index.

#### 5.1.4 Overview of Outcomes

Table 1 Primary and secondary outcomes

| | Data collection instrument and scale | Timepoints |
|---|---|---|
| rimary outcome | | |
| Probability of OMERACT-<br>OARSI response | The responder classification is a composite index reported as a single variable (yes/no) | t0, mo, t3, t6 |
| econdary outcomes | | |
| Hand pain at rest | Pain left/right hand last week, NRS 0-10, 0= no pain | t0, ex, mo, t3, t |
| Pain in activity | Pain left/right hand last week, NRS 0-10, 0= no pain | t0, ex, mo, t3, t |
| Stiffness | Stiffness left/right hand last week, NRS 0-10, 0= no stiffness | t0, ex, mo, t3, t |
| Grip strength | Maximum grip strength, mean of two measures left/right hand, in kg using the JAMAR dynamometer | t0, t3 |
| Activity performance of the hands (hand function) | Measured by the Measure of Activity Performance of the Hand (MAP-Hand); mean of 18 standardized activities, rating scale 1 ("no difficulty") to 4 ("cannot perform") | t0, mo, t3, t6 |
| Health-related quality of life | Measured by EuroQol EQ-5D-5L, five items (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) scored at a five level scare ("no problems" to "unable to do"), calculated as an utility index 0-1, 1= best health-related quality of life. Visual analogue scale (EQ VAS), 0-100, 100= perfect health | t0, t3, t6 |
| Global assessment of disease activity | Disease activity last week, NRS 0-10, 0=no disease activity | t0, mo, t3, t6 |
| Global assessment of change | 5-point Likert scale from "Much better" to "Much worse" | t3, t6 |
| Quality of care | Modified version of the OsteoArthritis Quality Indicator questionnaire, 15 questions rated as yes/no/unsure or not applicable, scored as pass rate 0-100, 100=best quality of care | t0, t3, t6 |
| Motivation for hand exercises | NRS 0-10, 10=highly motivated | t0, t3, t6 |

Statistical Analysis Plan Happy Hands Diakonhjemmet Hospital

Page 19 of 27

| | Hand exercises | Approximately number of exercise sessions each week for the last 3 months | t3, t6 |
|---|---|---|---|
| Cos | Costs | | |
| - | Healthcare use | Number of consultations with healthcare providers last 3 months | t3. t6 |
| | Medication use | Type and dosage last 3 months | t0, t3, t6 |
| | Hand surgery | Conducted hand surgery last 3 months (yes/no), if yes, reported sick leave due to hand surgery | t3, t6 |
| | Hospitalization | Number of hospital admissions | t3, t6 |
| | Medical equipment | Any medical equipment (i.e. hand orthoses, exercise equipment) bought last 3 months (type and cost) | t3, t6 |
| | Technical equipment | Any technical equipment (i.e. bread knife, jar key, sissors, electric toothbrush) bought last 3 months (type and cost) | t3, t6 |
| | Work status | Reported as yes/no on the following options: working, sick leave, retired, disability pension, work assessment allowance, unemployed, not working, student | t0, t3, t6 |
| Use | e <b>of the Happy Hands app</b> (inte<br>Usability | ervention group only) Measured by System Usability Scale (SUS), 10 statements scored on a 5-point scale from "strongly disagree" to "strongly agree" | t3, t6 |
| | Satisfaction with use of the app | NRS 0-10, 10=highly satisfied | t3, t6 |
| | Usefulness of the app | NRS 0-10, 10=highly useful | t3, t6 |
| | Adherence to hand | Number of exercises conducted | t3, (t6) |
| | exercises | | , , , |
| | Adherence to informational videos | Number of informational videos watched | t3, (t6) |
| | Adherence to guizzes | Number of quizzes answered | t3 |
| | Continued use | Plans to continue using the app, measured as yes/no/unsure | t3, t6 |
| | Adverse events | Description of any complaints related to hand exercises | t3 |
| , | | | ıs |
| Bas | seline characteristics | | |
| | Age | Years | t0 |
| | Gender | Female, male, other | t0 |
| | Living arrangement | Living alone, living together with someone | t0 |
| | Education | Elementary school, high school, university/college <4 years, university/college ≥ 4 years | t0 |
| | Smoking | No, previously, yes | t0 |
| | Height | Cm | t0 |
| | Weight | | t0 |
| | Most troublesome hand | Kg | |
| | | Left, right, both | t0 |
| | Other painful joints | Hip, knee, foot/ankle | t0 |
| | Previous treatment for HOA | Yes, no | t0 |
| | Previous hand surgery Comorbidities | Yes, no | t0 |
| | | High blood pressure, heart disease, lung disease, allergy, back pain, stroke, cancer, neurological disease, diabetes, metabolic | |
| | | disease, mental disease, kidney disease, liver disease, ulcer, blood disease | t0 |

Statistical Analysis Plan Happy Hands Diakonhjemmet Hospital

Health Literacy eHEALS, 5-point scale with a total score ranging from 8 to 40

(higher score representing higher health literacy) t0
Experience with using

technology and digital services

Experience with smartphone, tablets, apps, video consultation, and digital services (Helsenorge.no), measured on a 5-point scale (very poorly to very good) with an additional alternative of

'never tried' t0

Motivation for digital treatment/follow-up

reatment/follow-up NRS 0-10, 10=to a large degree t0

t0=baseline; t3=3 months; t6=6 months; ex=after each exercise session (in the app/intervention group only); mo=monthly (in the app/intervention group only); NRS=numeric rating scale; MAP-Hand=Measure of Activity Performance of the Hand; HOA=hand osteoarthritis

# 5.2 Analysis Methods

## 5.2.1 Primary Outcome

# 5.2.1.1 Primary Analysis

For analysis of the primary outcome a logistic regression with group as independent variable and OMERACT/OARSI response (yes/no) at 3 months as dependent variable will be conducted. The analysis will adjust for study center, the stratification factor used in the randomization. Probability of being a responder as well as risk difference will be calculated using the adjusted risk and risk difference estimators [25].

### 5.2.1.2 Additional analysis

Besides sensitivity analyses, no additional analyses are planned.

## 5.2.1.3 Summary Measures

See 5.1.1

## 5.2.1.4 Assumption Checks and Alternative Analyses

A logistic regression includes the following assumptions:

- Binary dependent variable: This assumption is fulfilled trough the study design. (OMERACT/OARSI responder criteria, calculated into a binary yes or no score).
- Independence: This assumption is fulfilled through the study design.
- No severe multicollinearity: This assumption is fulfilled through the study design.
- Sufficient number of observations: The sample size was calculated based on approximately 20% responders in the control group and 40% responders in the intervention group, which would provide sufficient number of patients per group.

# 5.2.1.5 Missing Data

We are expecting the amount of missing data to increase with time, but we cannot retrace the individual reasons for missingness. The primary analysis will utilize multiple imputation, including variables such as gender, age, pain, function and disease activity at baseline and 3 months.

# 5.2.1.6 Sensitivity Analyses

Statistical Analysis Plan Happy Hands Diakonhjemmet Hospital **Kommentert [JS1]:** Skal center justeres for? Vanlig å justere for stratifiseringsvariabler brukt i randomiseringen.

Page 21 of 27

For the primary endpoint, a sensitivity analysis will be carried out adjusting for recruitment site (, baseline pain, disease activity and function (which are the measures included in the OMERACT/OARSI responder criteria). Additional sensitivity analyses may be conducted, adjusting for variety in usual care (participating in osteoarthritis courses).

If deemed necessary, sensitivity analyses will also be conducted to address missing data and subgroup data.

## 5.2.1.7 Subgroup Analyses

No subgroup analyses are planned outside of the sensitivity analyses.

#### 5.2.2 Secondary Outcomes

## 5.2.2.1 Secondary Analyses

### a) OMERACT/OARSI responders at 6 months

For the secondary outcome of probability of OMERACT/OARSI response in the two groups at 6 months, we will conduct the same analysis as for the primary outcome.

Secondary continuous outcomes will be analysed using linear regression. The analyses will, in addition to randomization group, adjust for baseline level of the outcome and study center. Missing values will be handled using multiple imputation.

### b) Health economic evaluation

**Aim:** To assess whether the Happy Hands app in combination with usual care is a cost-effective treatment strategy for patients with hand OA compared to usual care alone.

**Statistical software:** Mainly STATA. Excel for bootstrap, plotting results on the cost-effectiveness plane and for construction the cost-effectiveness acceptability curve.

**Perspective on costs:** health care perspective as primary analysis, inclusion of production loss in explorative analysis.

**Cost of the intervention:** The Happy Hands app is not yet commercially available, hence has no official list price or yearly fee. Based on the cost of development and maintenance and the size of the eligible patient population, we assume that the app will be offered at an annual subscription fee of NOK 150 (EUR 13).

**Identification of resources:** patient self-reported in questionnaire, asked about resource use items as displayed in Table 1.

**Measurement of resource use:** patient self-reported in questionnaire. May add information from clinical expertise if needed, e.g. patient reports a rehabilitation stay, but not duration.

Valuation of resource use data: As far as possible, we will use unit prices reported in the Directorate of Medical Products database for use in health technology assessments (<a href="https://view.officeapps.live.com/op/view.aspx?src=https%3A%2F%2Fwww.dmp.no%2Fglobalassets%2Fdocuments%2Foffentlig-finansiering-og-pris%2Fdokumentasjon-til-metodevurdering%2Fenhetskostnader-v1.5.xlsx&wdOrigin=BROWSELINK), this includes the price per in-patient day at hospital.

If some unit price is not available in this database, we will use publicly available reimbursement rates. For visits to an occupational therapist in primary care, we will assume an average duration of visit and wage of therapist. Medical and technical equipment, such as a bread knife or vegetable knife with built-up handles, key for opening jars, or self-opening scissors, will be based on market prices (e.g. <a href="https://www.velferdsbutikken.no/categories/hielpemidler-kjokken">https://www.velferdsbutikken.no/categories/hielpemidler-kjokken</a>).

Identification of outcomes: self-reported in questionnaires.

**Measurement of outcomes:** Health related quality of life measured by the EQ-5D-5L. In the analysis of EQ-5D-5L, we will adjust for baseline imbalances using the method recommended by Manca and co-workers [26], if warranted.

**Valuation of outcomes:** Primary analysis based on the Norwegian EQ-5D-5L tariff by Garratt and cocorkers [27], sensitivity analysis with the UK Devlin tariff [28].

Analysis population: primary analysis with ITT population, may explore PP as sensitivity analysis.

**Timing:** Health-related quality of life is measured at baseline, 3 and 6 months, while costs are measured at 3 and 6 months.

Discounting: not relevant due to trial duration

**Cost-effectiveness threshold:** threshold suggested for Norway at time of analysis, currently NOK, 275,000 per QALY for patients with osteoarthritis

**Statistical decision rule:** Cost-effective if incremental cost-effectiveness ratio below threshold and if intervention has a higher probability of being cost-effective than comparator based on bootstrap results.

Analysis of resource use: mean cost per patient reported in 2024 EUR, will use valuta converter provided by "Norges Bank" to convert NOK to EUR using the average exchange rate in 2024 (https://www.norges-bank.no/tema/Statistikk/valutakurser/?tab=currency&frequencyTab=3).

Analysis of outcomes: mean QALY per patient. We expect no effect on mortality, hence any QALY gain will be a result of improvements in function and well-being. QALYs will be calculated based on the area under the curve approach. We will assume that transition between different health utility values will take place halfway between two measurements.

**Missing data:** if whole questionnaire of EQ-5D-5L is missing, multiple imputation, if single questions are missing, simple imputation. Costs are assumed to be missing only if the whole questionnaire is missing, if the questionnaire is missing, we will impute using multiple imputation.

Statistical Analysis Plan Happy Hands Diakonhjemmet Hospital

Analysis of cost-effectiveness: ICER=difference in mean costs/difference in mean QALY

Sampling uncertainty: We will use non-parametric bootstrapping to assess the degree of uncertainty around the ICER. We bootstrap costs and QALY 10,000 times with replacement, recalculate ICERS and plot the results on the cost-effectiveness plane. The likelihood of cost-effectiveness will then be calculated as the proportion of all bootstrapped samples below the cost-effectiveness threshold value. A cost-effectiveness acceptability curve will be constructed to illustrate how sensitive the conclusion is to varying levels of threshold values. This approach is one of several alternatives recommended for trial-based cost-effectiveness analyses [16].

Subgroup analysis: Per protocol population

Sensitivity analysis: Devlin tariff for the EQ-5D-5L

Explorative analysis: including loss of production

c) Effect on secondary outcomes (pain, hand function, grip strength, disease activity and quality of care)

To assess the effect of using the Happy Hands app in addition to usual care compared to usual care only on secondary outcomes of pain, hand function, grip strength, disease activity and quality of care, we will use multiple linear regression with the mean change scores at 3 and 6 months as dependent variables and group as independent variable, adjusting for baseline values for the variable of interest and recruitment sites.

## 5.2.2.2 Summary Measures

See 5.1.1

#### 5.2.2.3 Assumption Checks

A logistic regression includes the following assumptions:

- Binary dependent variable: This assumption is fulfilled trough the study design.
   OMERACT/OARSI responder criteria, calculated into a binary yes or no score.
- Independence: This assumption is fulfilled through the study design.
- No severe multicollinearity: This assumption is fulfilled through the study design.
- Sufficient number of observations: The sample size was calculated based on approximately 20% responders in the control group and 40% responders in the intervention group, which would provide sufficient number of patients per group.

A linear regression includes the following assumptions:

- Continuous dependent variable: This assumption is fulfilled through the study design.
- Independence: This assumption is fulfilled through the study design.
- Homoscedasticity: The spread of the residuals should be roughly the same across the regression line and should rather not exceed +3 and -3.

•

• Multicollinearity: The independent variables should not be highly correlated (r<0.7)

In case the outcome variable or the residuals are severly skewed, transformation (eg log-transformation) of the outcome variable will be carried out.

#### 5.2.2.4 Missing Data

We are expecting the amount of missing data to increase with time, but we cannot retrace the individual reasons for missingness. The cost-effectiveness analysis will utilize multiple imputation for missing whole questionnaires of EQ-5D. Costs will be assumed to be missing if the whole questionnaire is missing. If the questionnaire is answered without reporting costs, it will be assumed that the costs are 0. The other secondary analyses will be based on complete case analysis.

#### 5.2.2.5 Sensitivity Analyses

If deemed necessary, sensitivity analyses will also be conducted to address missing data and subgroup data.

#### 5.2.2.6 Subgroup Analyses

No subgroup analyses are planned outside of the sensitivity analyses.

### 5.2.3 Additional Analyses

#### 5.2.3.1 Exploratory Analyses

The following additional, hypothesis-generating, exploratory analyses will be conducted in addition to the above-stated analyses. If additional questions/analyses are raised during the analysis process, we will add them to this list of exploratory analyses.

- a) To assess the adherence, satisfaction and usability with use of the Happy Hands app, we will only include participants allocated to the intervention group. Adherence will be described with mean and SD or median and interquartile range, as well as the proportion of participants with adequate adherence to the exercise sessions and the information videos. Satisfaction and usability will be described with mean and SD or median and interquartile
- b) To identify relevant factors associated with being an OMERACT/OARSI responder at 3 and 6 months we will use multiple logistic regression and select variables based previous research and clinical relevance.
- c) To identify factors associated with adherence to the interventions (exercise and information videos) in the Happy Hands app, both multiple linear and logistic regression may be used.

# 6. Safety Analyses

## 6.1 Adverse Events/Safety

AEs is based on self-report in open-ended questions in the 3-months follow-up questionnaire and e-mails or phone calls from patients and will be categorised as mild to moderate depending on the

description in the questionnaire. Brief transitory pain/discomfort will be regarded as mild AEs and persistent pain/discomfort will be considered moderate AEs.

Per definition, any events caused by the intervention that results in significant disability, prolonged hospitalization, life threatening events or death are categorized as serious adverse events (SAE). As we did not expect that the intervention would cause any SAEs, we did not ask the patients for permission to retrieve information from their medical journal. Thus, information on life threatening events or death are not included in the study. Participants were asked about surgery and hospitalization due to hand osteoarthritis, however, planned surgery will not be considered an AE/SAE as this may be part of the treatment for these patients.

## 7. Statistical Software

All data handling and statistical analyses will be performed using Stata (StataCorp. 2015. College Station, TX, USA).

## 8. Ethics

The project is granted approval by the Regional Committees for Medical and Health Research Ethics (REK) in Norway (REK no 477746)

The study is funded by the Dam Foundation (2022/F0387170). The funders have no role in the study other than providing funding.

Data is stored in Services for sensitive data (TSD) at the University of Oslo and in a secure research server at Diakonhjemmet Hospital.

# 9. References

- 1. Cross M, Smith E, Hoy D, et al. (2014) The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Annals of the rheumatic diseases 73:1323-30. <a href="https://doi.org/10.1136/annrheumdis-2013-204763">https://doi.org/10.1136/annrheumdis-2013-204763</a>
- 2. Marshall M, Watt FE, Vincent TL, Dziedzic K (2018) Hand osteoarthritis: clinical phenotypes, molecular mechanisms and disease management. Nat Rev Rheumatol 14:641-56. <a href="https://doi.org/10.1038/s41584-018-0095-4">https://doi.org/10.1038/s41584-018-0095-4</a>
- 3. Qin J, Barbour KE, Murphy LB, et al. (2017) Lifetime Risk of Symptomatic Hand Osteoarthritis: The Johnston County Osteoarthritis Project. Arthritis Rheumatol 69:1204-12. https://doi.org/10.1002/art.40097
- 4. Kloppenburg M, Kroon FP, Blanco FJ, et al. (2018) 2018 update of the EULAR recommendations for the management of hand osteoarthritis. Ann Rheum Dis <a href="https://doi.org/10.1136/annrheumdis-2018-213826">https://doi.org/10.1136/annrheumdis-2018-213826</a>
- 5. Dziedzic KS, Allen KD (2018) Challenges and controversies of complex interventions in osteoarthritis management: recognizing inappropriate and discordant care. Rheumatology (Oxford, England) 57:iv88-iv98. <a href="https://doi.org/10.1093/rheumatology/key062">https://doi.org/10.1093/rheumatology/key062</a>
- $\label{eq:continuous} Kloppenburg M (2014) \ Hand \ osteoarthritis-nonpharmacological \ and \ pharmacological \ treatments. \ Nature \ reviews \ Rheumatology \ 10:242-51. \ \frac{https://doi.org/10.1038/nrrheum.2013.214}{https://doi.org/10.1038/nrrheum.2013.214}$

- 7. Gravås EMH, Tveter AT, Nossum R, et al. (2019) Non-pharmacological treatment gap preceding surgical consultation in thumb carpometacarpal osteoarthritis a cross-sectional study. BMC Musculoskelet Disord 20:180. https://doi.org/10.1186/s12891-019-2567-3
- 8. Ministry of Health and Care Services. [Meld. St. 9 Nasjonal helse- og samhandlingsplan 2024-2027 Vår felles helsetjeneste]. 2023-2024
- 9. Walter MM, Sirard P, Nero H, et al. (2023) Digitally delivered education and exercises for patients with hand osteoarthritis-An observational study. Musculoskeletal Care 21:1154-60. https://doi.org/10.1002/msc.1796
- Kroon FPB, Carmona L, Schoones JW, Kloppenburg M (2018) Efficacy and safety of non-pharmacological, pharmacological and surgical treatment for hand osteoarthritis: a systematic literature review informing the 2018 update of the EULAR recommendations for the management of hand osteoarthritis. RMD Open 4: https://doi.org/10.1136/rmdopen-2018-000734
- 11. Tveter AT, Varsi C, Maarnes MK, et al. (2024) Development of the Happy Hands selv-management app for people with hand osteoarthritits: a feasibility study. JMIR Form Res Sept 3 <a href="https://doi.org/10.2196/59016">https://doi.org/10.2196/59016</a>. [Epub ahead of print]
- 12. Tveter AT, Varsi C, Maarnes MK, et al. (2024) Development of the Happy Hands Self-Management App for People with Hand Osteoarthritis: Feasibility Study. JMIR Form Res 8:e59016. https://doi.org/10.2196/59016
- 13. Hennig T, Haehre L, Hornburg VT, Mowinckel P, Norli ES, Kjeken I (2015) Effect of home-based hand exercises in women with hand osteoarthritis: a randomised controlled trial. Annals of the rheumatic diseases 74:1501-8. https://doi.org/10.1136/annrheumdis-2013-204808
- 14. Østerås N, Hagen KB, Grotle M, Sand-Svartrud AL, Mowinckel P, Kjeken I (2014) Limited effects of exercises in people with hand osteoarthritis: results from a randomized controlled trial. Osteoarthritis and cartilage 22:1224-33. https://doi.org/10.1016/j.joca.2014.06.036
- 15. Dziedzic KS, Hill S, Nicholls E, et al. (2011) Self management, joint protection and exercises in hand osteoarthritis: a randomised controlled trial with cost effectiveness analyses. BMC musculoskeletal disorders 12:156. https://doi.org/10.1186/1471-2474-12-156
- 16. Ramsey SD, Willke RJ, Glick H, et al. (2015) Cost-effectiveness analysis alongside clinical trials II-An ISPOR Good Research Practices Task Force report. Value Health 18:161-72. https://doi.org/10.1016/j.jval.2015.02.001
- 17. Garber CE, Blissmer B, Deschenes MR, et al. (2011) American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc 43:1334-59. <a href="https://doi.org/10.1249/MSS.0b013e318213fefb">https://doi.org/10.1249/MSS.0b013e318213fefb</a>
- 18. Tveter AT, Østerås N, Nossum R, et al. (2020) Short-term effects of occupational therapy on hand function and pain in patients with carpometacarpal osteoarthritis: secondary analyses from a randomized controlled trial. Arthritis care & research https://doi.org/10.1002/acr.24543
- 19. Brørs G, Wentzel-Larsen T, Dalen H, et al. (2020) Psychometric Properties of the Norwegian Version of the Electronic Health Literacy Scale (eHEALS) Among Patients After Percutaneous Coronary Intervention: Cross-Sectional Validation Study. J Med Internet Res 22:e17312. <a href="https://doi.org/10.2196/17312">https://doi.org/10.2196/17312</a>
- 20. Norman CD, Skinner HA (2006) eHEALS: The eHealth Literacy Scale. J Med Internet Res 8:e27. https://doi.org/10.2196/imir.8.4.e27
- 21. Tveter AT, Nossum R, Eide REM, et al. (2020) The Measure of Activity Performance of the Hand (MAP-Hand) a reliable and valid questionnaire for use in patient with hand osteoarthritis with specific involvement of the thumb. J Hand Ther Submitted 28th October 2019:
- 22. Østerås N, Tveter AT, Garratt AM, et al. (2018) Measurement properties for the revised patient-reported OsteoArthritis Quality Indicator questionnaire. Osteoarthritis and cartilage 26:1300-10. <a href="https://doi.org/10.1016/j.joca.2018.06.007">https://doi.org/10.1016/j.joca.2018.06.007</a>
- 23. Herdman M, Gudex C, Lloyd A, et al. (2011) Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res 20:1727-36. https://doi.org/10.1007/s11136-011-9903-x
- 24. Pham T, van der Heijde D, Altman RD, et al. (2004) OMERACT-OARSI initiative: Osteoarthritis Research Society International set of responder criteria for osteoarthritis clinical trials revisited. Osteoarthritis and cartilage 12:389-99. https://doi.org/10.1016/j.ioca.2004.02.001
- 25. Kleinman LC, Norton EC (2009) What's the Risk? A simple approach for estimating adjusted risk measures from nonlinear models including logistic regression. Health Serv Res 44:288-302. https://doi.org/10.1111/j.1475-6773.2008.00900.x
- 26. Manca A, Hawkins N, Sculpher MJ (2005) Estimating mean QALYs in trial-based cost-effectiveness analysis: the importance of controlling for baseline utility. Health Econ 14:487-96. https://doi.org/10.1002/hec.944
- 27. Garratt AM, Stavem K, Shaw JW, Rand K (2025) EQ-5D-5L value set for Norway: a hybrid model using cTTO and DCE data. Qual Life Res 34:417-27. https://doi.org/10.1007/s11136-024-03837-3
- 28. Devlin NJ, Shah KK, Feng Y, Mulhern B, van Hout B (2018) Valuing health-related quality of life: An EQ-5D-5L value set for England. Health Econ 27:7-22. <a href="https://doi.org/10.1002/hec.3564">https://doi.org/10.1002/hec.3564</a>